CLINICAL TRIAL: NCT00670553
Title: A Phase I Study of LBH589 (Panobinostat) in Combination With External Beam Radiotherapy for the Treatment of Prostate Cancer, Esophageal Cancer and Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589CBE01
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer; Head & Neck Cancer; Esophageal Cancer
Keywords: Prostate,; Head & Neck,; Esophageal
MeSH Terms: conditions — Prostatic Neoplasms; Head and Neck Neoplasms; Esophageal Neoplasms | interventions — Panobinostat

ARMS (1):
- LBH589 (Experimental)
  Interventions: Drug: panobinostat

INTERVENTIONS:
Drug: panobinostat
  Other Names: LBH589

SUMMARY:
The purpose of this study is to assess the feasibility of combined administration of different LBH589 dosages with radiotherapy in order to establish the dosage to be evaluated in future studies.

ELIGIBILITY:
Inclusion criteria:

* Patients with age ≥18 years
* Confirmed diagnosis of prostate cancer, SCC esophageal cancer or head & neck cancer
* No evidence of distant spread of the disease

Exclusion criteria:

* Patients who have severe and/or uncontrolled medical conditions
* Female patients who are pregnant or breast feeding

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Establish Dose Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD) | 1 to 28 days

SECONDARY OUTCOMES:
Safety profile of oral LBH589 when given in combination with standard Radiotherapy | min 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Liège, Belgium